CLINICAL TRIAL: NCT05526742
Title: A Randomized, Open-Label, Crossover Study to Evaluate the Relative Bioavailability of a Tablet Formulation of CKD-510 as Compared to Capsule and to Assess the Effect of Food on the CKD 510 Tablet Formulation in Healthy Subjects
Brief Title: A Study to Evaluate the Relative Bioavailability of Formulations of CKD-510 and to Assess the Effect of Food on the CKD-510 Tablet Formulation in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A96_03PK2212
Record Dates: First submitted 2022-08-31; First posted 2022-09-02 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Subjects will receive single-dose of CKD-510 capsule in fasted state (treatment A) on Day 1 of Period 1 and tablet in fasted state (treatment B) on Day 1 of Period 2, and then receive tablet in a fed state (treatment C) on Day 1 of Period 3.
  A washout period will be at least 7 days between each treatment period.
  Interventions: Drug: CKD-510 capsule (reference); Drug: CKD-510 tablet (test)
- Group 2 (Experimental): Subjects will receive single-dose of CKD-510 tablet in a fed state (treatment C) on Day 1 of Period 1 and tablet in fasted state (treatment B) on Day 1 of Period 2, and then receive capsule in fasted state (treatment A) on Day 1 of Period 3.
  A washout period will be at least 7 days between each treatment period.
  Interventions: Drug: CKD-510 capsule (reference); Drug: CKD-510 tablet (test)

INTERVENTIONS:
Drug: CKD-510 capsule (reference) — Single-dose of CKD-510 will be administered as oral capsule in a fasted state.
Drug: CKD-510 tablet (test) — Single-dose of CKD-510 will be administered as oral tablet in a fasted state.
Drug: CKD-510 tablet (test) — Single-dose of CKD-510 will be administered as oral tablet in a fed state.

SUMMARY:
The purpose of this study is to determine the relative bioavailability of CKD-510 tablet formulation compared with CKD-510 capsule formulation, and to characterize the effect of food on the CKD-510 tablet.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male or female subject between 18 and 60 years of age
* In generally good health, based upon medical/surgical history and the results of physical examination, vital signs, safety laboratory assessments, and 12-lead ECG
* Body mass index (BMI) between 18 and 32 kg/m2
* If a female subject of childbearing potential, agrees to use a highly effective method of contraception during study participation and for 90 days after the last administration of study drug.
* If a male subject with a female partner of childbearing potential, is surgically sterile or agrees to use a highly effective method of contraception during study participation and for 90 days after the last administration of study drug
* Negative test result for SARS-CoV-2

Exclusion Criteria:

* Evidence of clinically significant hematologic, renal, endocrine, pulmonary, cardiac, gastrointestinal, hepatic, psychiatric, neurologic, immunologic, or allergic disease or any other condition
* Any hypersensitivity or allergy to CKD-510 or its excipients or to any medicinal products with similar chemical structures
* History of malignancy, other than successfully treated basal cell or squamous cell skin cancer
* History or presence of an abnormal 12-lead ECG
* Acute illness considered clinically significant by the Investigator within 30 days prior to Randomization
* Any other investigational drug within 30 days or 5 half-lives of the drug (whichever is longer) prior to Randomization

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2022-08-24 (Actual); Primary Completion 2022-09-13 (Actual); Study Completion 2022-09-13 (Actual)

PRIMARY OUTCOMES:
Plasma Cmax after administration of either capsule or tablet formulation in fasted state | From Day 1 to Day 3 of each Treatment Period
  Maximum plasma concentration (Cmax)
Plasma AUC after administration of either capsule or tablet formulation in fasted state | From Day 1 to Day 3 of each Treatment Period
  Area under the concentration-time curve (AUC)
Plasma Tmax after administration of either capsule or tablet formulation in fasted state | From Day 1 to Day 3 of each Treatment Period
  Time to maximum plasma concentration (Tmax)
Plasma T1/2 after administration of either capsule or tablet formulation in fasted state: T1/2 | From Day 1 to Day 3 of each Treatment Period
  Terminal phase elimination half-life (T1/2)
Plasma Cmax after administration of tablet formulation in the fed and fasted states | From Day 1 to Day 3 of each Treatment Period
  Maximum plasma concentration (Cmax)
Plasma AUC after administration of tablet formulation in the fed and fasted states | From Day 1 to Day 3 of each Treatment Period
  Area under the concentration-time curve (AUC)
Plasma Tmax after administration of tablet formulation in the fed and fasted states | From Day 1 to Day 3 of each Treatment Period
  Time to maximum plasma concentration (Tmax)
Plasma T1/2 after administration of tablet formulation in the fed and fasted states | From Day 1 to Day 3 of each Treatment Period
  Terminal phase elimination half-life (T1/2)
Safety and tolerability including treatment-emergent AE and treatment-emergent SAE | From Day 1 to Day 7

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Pharmacology Unit, Cincinnati, Ohio, United States